CLINICAL TRIAL: NCT00068653
Title: Phase II Study of the Combination of ZD1839 (Iressa) and Celecoxib in Patients With Platinum Refractory Non-Small Cell Lung Cance
Brief Title: Gefitinib and Celecoxib in Treating Patients With Refractory Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000327805; P30CA022453 (NIH); WSU-C-2563; ZENECA-1839US/0252
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Celecoxib & ZD1839 (Experimental): Celecoxib: 400mg orally two times a day, taken with meals.
  ZD1839: 250 mg po every day, taken with or without food.
  Interventions: Drug: Celecoxib; Drug: ZD1839

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 400mg orally two times a day, taken with meals.
  Other Names: Celebrex
Drug: ZD1839 — ZD1839 250 mg po every day, taken with or without food.
  Other Names: Iressa; Gefitinib

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Celecoxib may slow the growth of cancer by stopping blood flow to the tumor. Combining gefitinib with celecoxib may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gefitinib with celecoxib in treating patients who have non-small cell lung cancer that is refractory to platinum-based chemotherapy (such as cisplatin or carboplatin).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with platinum-refractory non-small cell lung cancer treated with gefitinib and celecoxib.

Secondary

* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive oral gefitinib once daily and oral celecoxib twice daily on days 1-28. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for up to 6 weeks.

PROJECTED ACCRUAL: A total of 18-27 patients will be accrued for this study within 22 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)
* Progression of disease during platinum-based (cisplatin or carboplatin) chemotherapy or within 3 months of completing chemotherapy

  * Treatment with other agents since prior platinum-based chemotherapy allowed
* Measurable disease

  * Target lesions within a prior radiation field must have documented evidence of progression at least 8 weeks after the completion of radiotherapy
* No active brain or leptomeningeal metastases

  * Treated brain metastases allowed at least 4 weeks after the completion of appropriate therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN (if alkaline phosphatase is no greater than ULN)
* Alkaline phosphatase no greater than 5 times ULN (if AST and ALT are greater than ULN)
* No history of chronic hepatitis

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No active thromboembolic event within the past 4 weeks
* No uncontrolled congestive heart failure
* No uncontrolled angina
* No myocardial infarction and/or stroke within the past 6 months

Pulmonary

* No evidence of clinically active interstitial lung disease

Gastrointestinal

* No history of gastrointestinal bleeding within the past 6 months
* No history of peptic ulcer disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must weigh at least 110 pounds (50 kg)
* HIV negative
* No allergy to sulfonamides
* No allergy to any NSAID, including celecoxib
* No known severe hypersensitivity to gefitinib or any of its excipients
* No other malignancy within the past 3 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No history of dementia, active psychiatric disorder, or any other condition that would preclude study compliance
* No other concurrent serious medical condition

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior epidermal growth factor receptor inhibitor
* No concurrent biologic therapy

Chemotherapy

* See Disease Characteristics
* More than 2 weeks since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Recovered from prior radiotherapy

Surgery

* Recovered from prior surgery

Other

* Recovered from prior therapy
* More than 2 weeks since prior investigational therapy
* More than 1 week since prior fluconazole
* More than 30 days since prior participation in another investigational agent clinical trial
* More than 30 days since prior chronic nonsteroidal anti-inflammatory drugs (NSAIDs), including celecoxib or rofecoxib
* No prior gefitinib
* No prior cyclooxygenase-2 (COX-2) inhibitor or another clinical trial for NSCLC
* No other concurrent NSAIDs

  * Concurrent aspirin allowed (not to exceed 325 mg/day)
* No other concurrent COX-2 inhibitors
* No concurrent lithium
* No concurrent fluconazole
* No concurrent use of any of the following:

  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Rifampin
  * Phenobarbital
  * Hypericum perforatum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-06; Primary Completion 2007-10 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Response rate | Every 2 cycles; after the 1st 4 cycles, every month by clinical exam & every 3 months radiological evaluation
  CT scan chest/abdomen; Assessments of complete response (CR) or partial response (PR)require confirmation 4 weeks or later.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Every 2 cycles; after the 1st 4 cycles, every month by clinical exam & every 3 months radiological evaluation
Overall survival | Every 2 cycles; after the 1st 4 cycles, every month by clinical exam & every 3 months radiological evaluation
Toxicity of this drug combination | Every 2 weeks; Every month after 4 cycles if the patient has not developed > Grade 2 toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M. Gadgeel, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States